CLINICAL TRIAL: NCT03349814
Title: Explanations for Negative Laparoscopic Appendectomies and Normal Laparoscopies. What Does the Patient Suffer From When the Appendix Proves to be Healthy?
Brief Title: Explanations for Negative Laparoscopic Appendectomies and Normal Laparoscopies
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Siv Fonnes, MD, PhD-student, Herlev Hospital
Other Study IDs: HEH-TR-1
Record Dates: First submitted 2017-11-01; First posted 2017-11-22 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Appendicitis; Yersinia Enterocolitica Infection; Yersinia Pseudotuberculosis Infections; Appendectomy
Keywords: appendicitis; appendectomy; yersinia
MeSH Terms: conditions — Appendicitis; Yersinia Infections; Yersinia pseudotuberculosis Infections | interventions — Laparoscopy; Appendectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serology samples: collected for the current research project, analyzed at Statens Serum Institut (SSI), and thereafter anonymized and transferred to the biobank of SSI.
  EDTA-blood samples, serum-blood samples and buffycoat: collected only for the biobank for future research. Stored for 10 years at Herlev Hospital, and thereafter destroyed.
  Rectal swab: collected for the current research project. Appendix swab: collected only for the biobank for future research. Stored at Herlev Hospital in the biobank for future research for 10 years, thereafter destroyed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Appendicitis group: Patients, who undergo a diagnostic laparoscopy, which because of the operative findings leads to an appendectomy, and the appendix is found to be inflamed in the pathology report.
  A diagnostic laparoscopy where the appendix seems inflamed, and therefore is removed.
  Interventions: Procedure: Diagnostic laparoscopy with appendectomy
- Normal appendix group: Patients, who undergo a diagnostic laparoscopy, that either because of the operative findings (mesenteric lymphadenitis or normal diagnostic laparoscopy) does not lead to appendectomy, or leads to appendectomy, but the appendix is not found to be inflamed in the pathology report.
  A diagnostic laparoscopy where the appendix is not found to be inflamed, and therefore is not removed.
  OR
  A diagnostic laparoscopy where the appendix seems inflamed, and therefore is removed, but is not found to be inflamed in the pathology report.
  Interventions: Procedure: Diagnostic laparoscopy without appendectomy; Procedure: Diagnostic laparoscopy with appendectomy

INTERVENTIONS:
Procedure: Diagnostic laparoscopy without appendectomy — A diagnostic laparoscopy where the appendix is not found to be inflamed, and therefore is not removed.
  Groups: Normal appendix group
Procedure: Diagnostic laparoscopy with appendectomy — A diagnostic laparoscopy where the appendix seems inflamed, and therefore is removed

SUMMARY:
Trial The aim of the study is to investigate which infectious diseases might mimic the symptoms of acute appendicitis to a degree to cause a diagnostic laparoscopy or laparoscopic appendectomy. The primary outcome is to compare the incidence of Yersinia spp. infection in patients, who undergo surgery due to suspected appendicitis, between those with and without appendicitis detected by polymerase chain reaction on rectal swabs. The secondary outcomes are comparison of the incidence of bacterial pathogens (Campylobacter spp., Salmonella spp., Shigella spp., Aeromonas spp.) and Enterobius vermicularis in the two groups. Rectal swabs, appendix swabs, and blood samples are collected prospectively and research biobanks will be established. Initially, the rectal samples and serology samples will be investigated, and possible biomarkers and results of the appendix swabs will be evaluated at a later time point.

Ethics The trial will be conducted according to the Helsinki II Declaration after approval from both the local Health Research Ethics Committee and the Danish Data Protection Agency. An informed written consent will be collected from the participants prior to inclusion in the study. Data will be stored according to the approval from the Danish Data Protection Agency. This study is conducted in patients with suspected appendicitis. These patients are fully awake and conscious at time of inclusion. The patients included in this study will not experience any adverse effects due to their participation.

DETAILED DESCRIPTION:
Aim The aim of the study is to investigate which infectious diseases might mimic the symptoms of acute appendicitis to a degree that cause a diagnostic laparoscopy or laparoscopic appendectomy.

Primary outcome A comparison of the incidence of Yersinia spp. (enterocolitica and/or pseudotuberculosis) infection diagnosed by PCR on rectal swabs in the two groups: patients with histopathological confirmed inflammation (appendicitis group) and patients with one of the following: a histopathological normal appendix without inflammation, mesenteric lymphadenitis, or a normal diagnostic laparoscopy (normal appendix group).

Secondary outcomes A comparison of the incidence of other microbes: Campylobacter spp., Salmonella spp., Shigella spp., and Aeromonas spp. found by PCR of rectal swabs in the two groups: normal appendix versus appendicitis group.

Patients positive for Yersinia spp. will be evaluated individually in subgroups of the two groups: appendicitis group and normal appendix group. Serological investigation for Yersinia will be conducted if funding is achieved.

A comparison of the incidence of Enterobius vermicularis found in the histopathological examination in the two groups.

Design A prospective, observational cohort study. Trial participants Inclusion criteria

* ≥18 years old
* Suspicion of acute appendicitis and planned for diagnostic laparoscopy
* Written informed consent after written and verbal information Exclusion criteria
* Cannot understand, read or speak Danish
* Known with inflammatory bowel disease
* Other intra-abdominal pathology than appendicitis requiring other surgical intervention or treatment (diagnosed either perioperatively, at a preoperative CT-scan, or shortly after the surgery in the histopathological examination)
* Not undergoing diagnostic laparoscopy, laparoscopic appendectomy, or open appendectomy
* Use of antimicrobial agents within two weeks prior to inclusion until actual admission for acute abdominal pain

Trial course Patients are admitted to the Department of Surgery, Herlev Hospital, with suspected acute appendicitis. A surgeon from the department will either plan for an acute surgery or keep patients for further observation. The investigators of the trial or research assistants will approach these patients to give information about the study. Thereby, the investigators ensure the patient has as much time as possible for consideration in this acute setting. Patients, who fulfill the inclusion criteria and none of the exclusion criteria (apart from those criteria that can only be clarified at or after surgery), are included in the trial after informed consent. Baseline characteristics of the enrolled patients including their medical history, travel history and gastrointestinal symptoms will be registered in the electronic case report forms (eCRF) in RedCAP. Blood samples and a rectal swab are collected before surgery. A note of the patient's inclusion in the trial will be added to the patient's medical record. Included patients will undergo a diagnostic laparoscopy performed according to standard clinical practice. If the appendix is removed during surgery, a swab from the removed appendix will be collected postoperatively. The appendix swab will only be collected if the appearance of the removed appendix is not suspicious for malignant disease (SOP_Appendixpodning). This is in agreement with the Department of Pathology, Herlev Hospital, not to compromise the histopathological examination and to prevent spread of malignant cells in the rare case of an appendix tumor. If there is any doubt regarding the appearance of the appendix no swab will be collected. A follow-up of the patient's medical record with regard to the pathology report will be conducted ten days after surgery. These results are noted in the patient's eCRF.

Withdrawal and drop-out criteria The participants can withdraw their consent at any point during the trial. The collected blood samples, rectal swab and possible appendix swab will be destroyed if a participant withdraws consent. A participant has concluded the trial ten days after surgery when both the final record of the surgery and pathology report is available. Patients, who during or shortly after surgery fulfill any exclusion criterion regarding other intra-abdominal pathology, conditions requiring other treatment, or do not undergo the planned surgery, will drop out of the study and will thus be excluded from the study and the collected blood sample, rectal swab, and possible appendix swab will be destroyed. A participant has concluded the study when the 10-day postoperative follow-up has been conducted.

Primary outcome

The primary outcome will be based on the cumulative results from both methods:

• Detection of infection with Yersinia spp. (enterocolitica and/or pseudotuberculosis) by microbiological investigation of rectal swab: Specimens (rectal swab) collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, a fraction of the collected specimens from each patient is sent to the Department of Clinical Microbiology, Hvidovre Hospital and thereafter investigated with a real time PCR for Yersinia spp. These results are noted in the patient's eCRF, but not in the patient's medical record. Samples with a positive PCR result will be cultured for Yersinia spp. and in case of positive culture results, susceptibility testing will be performed (secondary outcome). Hereafter, the collected human material and the cultured Yersinia enterocolitica will be frozen at -80°C and stored for ten years at Hvidovre Hospital as a biobank for future research.

Secondary outcomes

* Serology of Yersinia enterocolitica: This outcome will be reported on in the planned publication if sufficient funding is achieved, otherwise, it will be presented in a later publication. Six ml of blood collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, the blood sample for serology from each patient is sent to Statens Serum Institut. Here, the blood samples are investigated a soon as possible after arrival with an in-house ELISA test for Yersinia enterocolitica IgM, IgA, and IgG. After the analysis, the serum samples will be frozen at -80°C and stored for ten years at Statens Serum Institut as a biobank for future research. Thereafter, the samples will be anonymized and transferred to the biobank for future research belonging to Statens Serum Institut.
* Detection of other bacterial pathogens: The specimens (rectal swab) collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, a fraction of the collected specimens from each patient is sent to the Department of Clinical Microbiology, Hvidovre Hospital and thereafter investigated with a multiplex real time PCR for:

  * Campylobacter spp.
  * Salmonella spp.
  * Shigella spp.
  * Aeromonas spp. Samples with positive PCR results for bacterial pathogens will be cultured (including Yersinia spp.) and in case of positive culture, susceptibility testing will be performed. Hereafter, the collected human material and the cultured bacteria will be frozen at -80°C and stored for ten years at that site as a research biobank, hereafter samples are anonymized.
* Combined outcome of serology and PCR for Yersinia spp.: See description above. This outcome will only be reported if funding is achieved.
* Plasma and full blood are kept for later analysis. 12 ml of blood will be collected per patient: 6 ml will be used to make EDTA-plasma samples and buffycoat and 6 ml will be stored as serum samples. A research biobank will be established for the collected samples, which will be frozen and stored at -80°C for ten years. Thereafter the plasma and full blood samples are destroyed. The local Health Research Ethics Committee (Capital region of Denmark) will be contacted regarding the use of this research biobank before further investigations are initiated. The participants will be asked for consent specifically regarding the biological material for the biobank for future research.
* The remaining fractions of specimens from the rectal swabs and specimens from the appendix swabs are stored for later analysis. A research biobank will be established for the collected samples at Herlev Hospital, which will be frozen and stored at -80°C for ten years. Thereafter the specimens are destroyed. The local Health Research Ethics Committee (Capital region of Denmark) will be contacted regarding the use of the research biobank before further investigations are initiated. The participants will be asked for consent specifically regarding the biological material for the biobank for future research.

Statistics Continuous numerical data will be reported as mean and standard deviation if normally distributed. If not normally distributed, continuous numerical data will be reported as median and percentiles. The investigators will analyze data with both parametric and non-parametric statistics depending on the distribution of the data. A p-value <0.05 is considered significant.

The power calculation is as follows. The rate of Yersinia spp. in the appendicitis group is expected to be 13%. The sizes of the groups are expected to be unequal. Approximately 80% of the included patients will be in the appendicitis group and 20% will be in the normal appendix group.

When alfa is set at 0.05, beta is set at 0.80, and the least interesting difference between the groups is set at 20%, a total of 225 patients are required: 45 patients in the normal appendix group and 180 patients in the appendicitis group.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of acute appendicitis and planned for diagnostic laparoscopy
* Written informed consent after written and verbal information

Exclusion Criteria:

* Cannot understand, read or speak Danish
* Known with inflammatory bowel disease
* Other intra-abdominal pathology than appendicitis requiring other surgical intervention or treatment (diagnosed either perioperatively, at a preoperative CT-scan, or shortly after the surgery in the histopathological examination)
* Not undergoing diagnostic laparoscopy, laparoscopic appendectomy, or open appendectomy
* Use of antimicrobial agents within two weeks prior to inclusion until actual admission for acute abdominal pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult with suspection of acute appendicits can be included in the study, unless they have known inflammatory bowel disease or another intra-abdominal pathology that appendicitis.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-28 (Actual)

PRIMARY OUTCOMES:
Detection of infection with Yersinia spp. (enterocolitica and/or pseudotuberculosis) by microbiological investigation of rectal swab | We follow every patient from admission through surgery and until pathology report approximately ten days after surgery. The analyses are done after the last patient has concluded the trial. We expect the data collection process to take about a year.
  Specimens (rectal swab) collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, a fraction of the collected specimens from each patient is sent to the Department of Clinical Microbiology, Hvidovre Hospital and thereafter investigated with a real time PCR for Yersinia spp. These results are noted in the patient's eCRF, but not in the patient's medical record. Samples with a positive PCR result will be cultured for Yersinia spp. and in case of positive culture results, susceptibility testing will be performed (secondary outcome). Hereafter, the collected human material and the cultured Yersinia enterocolitica will be frozen at -80°C and stored for ten years at Hvidovre Hospital as a biobank for future research.

SECONDARY OUTCOMES:
Serology of Yersinia enterocolitica | We follow every patient from admission through surgery and until pathology report approximately ten days after surgery. The analyses are done after the last patient has concluded the trial. We expect the data collection process to take about a year.
  This outcome will be reported on in the planned publication if sufficient funding is achieved, otherwise, it will be presented in a later publication. Six ml of blood collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, the blood sample for serology from each patient is sent to Statens Serum Institut. Here, the blood samples are investigated a soon as possible after arrival with an in-house ELISA test for Yersinia enterocolitica IgM, IgA, and IgG. After the analysis, the serum samples will be frozen at -80°C and stored for ten years at Statens Serum Institut as a biobank for future research. Thereafter, the samples will be anonymized and transferred to the biobank for future research belonging to Statens Serum Institut.
Detection of infection with Yersinia spp. by either serology or PCR for Yersinia spp. | We follow every patient from admission through surgery and until pathology report approximately ten days after surgery. The analyses are done after the last patient has concluded the trial. We expect the data collection process to take about a year.
  See descriptions for outcome 1 and outcome 2. The overall prevalence of Yersinia spp. detected by either serology or PCR will be reported. This outcome will be based on the cumulative results from both methods. This outcome will only be reported if funding is achieved.
Detection of Campylobacter spp. | We follow every patient from admission through surgery and until pathology report approximately ten days after surgery. The analyses are done after the last patient has concluded the trial. We expect the data collection process to take about a year.
  The specimens (rectal swab) collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, a fraction of the collected specimens from each patient is sent to the Department of Clinical Microbiology, Hvidovre Hospital and thereafter investigated with a multiplex real time PCR for Campylobacter spp.
  Samples with positive PCR results for bacterial pathogens will be cultured (including Yersinia spp.) and in case of positive culture, susceptibility testing will be performed. Hereafter, the collected human material and the cultured bacteria will be frozen at -80°C and stored for ten years at that site as a research biobank, hereafter samples are anonymized.
Detection of Salmonella spp. | We follow every patient from admission through surgery and until pathology report approximately ten days after surgery. The analyses are done after the last patient has concluded the trial. We expect the data collection process to take about a year.
  The specimens (rectal swab) collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, a fraction of the collected specimens from each patient is sent to the Department of Clinical Microbiology, Hvidovre Hospital and thereafter investigated with a multiplex real time PCR for Salmonella spp.
  Samples with positive PCR results for bacterial pathogens will be cultured (including Yersinia spp.) and in case of positive culture, susceptibility testing will be performed. Hereafter, the collected human material and the cultured bacteria will be frozen at -80°C and stored for ten years at that site as a research biobank, hereafter samples are anonymized.
Detection of Shigella spp. | We follow every patient from admission through surgery and until pathology report approximately ten days after surgery. The analyses are done after the last patient has concluded the trial. We expect the data collection process to take about a year.
  The specimens (rectal swab) collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, a fraction of the collected specimens from each patient is sent to the Department of Clinical Microbiology, Hvidovre Hospital and thereafter investigated with a multiplex real time PCR for Shigella spp.
  Samples with positive PCR results for bacterial pathogens will be cultured (including Yersinia spp.) and in case of positive culture, susceptibility testing will be performed. Hereafter, the collected human material and the cultured bacteria will be frozen at -80°C and stored for ten years at that site as a research biobank, hereafter samples are anonymized.
Detection of Aeromonas spp. | We follow every patient from admission through surgery and until pathology report approximately ten days after surgery. The analyses are done after the last patient has concluded the trial. We expect the data collection process to take about a year.
  The specimens (rectal swab) collected prior to surgery are immediately frozen at -80°C and stored at Herlev Hospital in a research biobank. When the last patient has concluded the trial, a fraction of the collected specimens from each patient is sent to the Department of Clinical Microbiology, Hvidovre Hospital and thereafter investigated with a multiplex real time PCR for Aeromonas spp.
  Samples with positive PCR results for bacterial pathogens will be cultured (including Yersinia spp.) and in case of positive culture, susceptibility testing will be performed. Hereafter, the collected human material and the cultured bacteria will be frozen at -80°C and stored for ten years at that site as a research biobank, hereafter samples are anonymized.

CONTACTS AND LOCATIONS:
Overall Officials: Siv Fonnes, MD, Principal Investigator — Centre for Perioperative Optimization, Department of Surgery, Herlev and Gentofte Hospitals, University of Copenhagen
Locations (1):
- Herlev Hospital, Herlev, Capital Region of Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Humes DJ, Simpson J. Acute appendicitis. BMJ. 2006 Sep 9;333(7567):530-4. doi: 10.1136/bmj.38940.664363.AE. No abstract available. PMID 16960208
- [Background] Frisch M, Pedersen BV, Andersson RE. Appendicitis, mesenteric lymphadenitis, and subsequent risk of ulcerative colitis: cohort studies in Sweden and Denmark. BMJ. 2009 Mar 9;338:b716. doi: 10.1136/bmj.b716. PMID 19273506
- [Background] Slotboom T, Hamminga JT, Hofker HS, Heineman E, Haveman JW; Apple Study Group Appendicitis and Laparoscopic Evaluation. Intraoperative motive for performing a laparoscopic appendectomy on a postoperative histological proven normal appendix. Scand J Surg. 2014 Dec;103(4):245-8. doi: 10.1177/1457496913519771. Epub 2014 Apr 15. PMID 24737848
- [Derived] Fonnes S, Mollerup S, Paulsen SJ, Petersen AM, Holzknecht BJ, Westh H, Rosenberg J. A prospective cohort study of the rectal microbiome in patients with suspected appendicitis. Clin Res Hepatol Gastroenterol. 2025 Sep-Oct;49(8):102675. doi: 10.1016/j.clinre.2025.102675. Epub 2025 Aug 21. PMID 40848874
- [Derived] Fonnes S, Mollerup S, Paulsen SJ, Holzknecht BJ, Westh H, Rosenberg J. The microbiome of the appendix differs in patients with and without appendicitis: A prospective cohort study. Surgery. 2024 Jun;175(6):1482-1488. doi: 10.1016/j.surg.2024.02.020. Epub 2024 Apr 1. PMID 38565493